CLINICAL TRIAL: NCT02029313
Title: A Randomized, Open-label, Single-Dose, 2-Treatment, 2-Way, 2-Period Crossover Study to Compare the Safety and the Pharmacokinetic Characteristics of MKT-N2 (Montelukast) and Singulair® (Montelukast Sodium) Tablet 10mg in Healthy Male Korean Subjects
Brief Title: Safety and the Pharmacokinetic Study of Characteristics of MKT-N2 (Montelukast) and Singulair® (Montelukast Sodium)to Treat Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PMK-M01RS1
Record Dates: First submitted 2013-11-03; First posted 2014-01-07 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Asthma and Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MKT-N2 (Experimental): Montelukast
  Interventions: Drug: Montelukast; Drug: Montelukast sodium
- Singulair (Active Comparator): Montelukast sodium
  Interventions: Drug: Montelukast; Drug: Montelukast sodium

INTERVENTIONS:
Drug: Montelukast
Drug: Montelukast sodium

SUMMARY:
The Purpose of A center, Randomized, Open label, single dose, Placebo-controlled, 2-Treatment, 2-Way, 2-Period Crossover Study to Compare the Safety and the Pharmacokinetic Characteristics of MKT-N2 (Montelukast) and Singulair® (montelukast sodium) tablet 10mg in Healthy Male Korean Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Korean Male over20, under 45 years old
* 55kg over weight, IBW +-20% range male

Exclusion Criteria:

* Males who have gotten a clinically significant of liver, pancreas, kidneys, nervous system, respiratory system, endocrine system, blood cancer, mental illness, cardiovascular, urinary tract disease, or a history corresponding
* Males who have gotten a history of gastrointestinal disease
* Males who have gotten a history of hypersensitivity to montelukast or reaction to other drugs(aspirin, antibiotics)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse event | 1day

SECONDARY OUTCOMES:
Pharmacokinetic profiles | 1day
  Blood evaluation variables: Cmax, AUCt (t=24 h), AUC∞, tmax

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, Junggu, South Korea